CLINICAL TRIAL: NCT01128062
Title: Canthaxanthin Retinopathy: A Long-term Observation
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Other Study IDs: AHARMS-8310
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-05

CONDITIONS: Canthaxanthin Retinopathy
Keywords: Canthaxanthin retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Canthaxanthine is a naturally occurring carotenoid that has been a popular over-the-counter oral artificial tanning agent in Europe, Canada, and Australia since 1979. It is also used at low dosage as a food-colouring agent and as a therapeutic agent for photosensitivity disorders such as erythropoietic protoporphyria. Canthaxanthin retinopathy was first described in 1982 by Cortin et al. In Germany the office of the federal board of health refused the permit for oral tanning agents containing canthaxanthine in 1985. At that time the long-term course of the disease was not known. 25 years later the investigators did these long-term follow-up examinations.

ELIGIBILITY:
Inclusion Criteria:

* patients using oral tanning agents for at least 2 months.
* patients of 18 years or older

Exclusion Criteria:

* none.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of oral tanning agents should report at the University Eye hospital for examination.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 1983-12; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
all eye diseases | 2008 and 2009
  All patients will have the follow-up examination 2008 or 2009. The examination included at most visual acuity (distant and near vision), Amsler test, examination of anterior segment, posterior segment, 10-2 and 30-2 visual field, electrooculography, electroretinography, multifocal electroretinography, fundus photography, fluorescein angiography, and an examination for autofluorescence.

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, University of Cologne, Cologne, North Rhine-Westphalia, Germany